CLINICAL TRIAL: NCT03866239
Title: A Phase Ib, Multicenter, Open-Label Study to Evaluate the Safety, Efficacy, and Pharmacokinetics of Cibisatamab in Combination With Atezolizumab After Pretreatment With Obinutuzumab in Patients With Previously Treated Metastatic, Microsatellite-Stable Colorectal Adenocarcinoma With High CEACAM5 Expression
Brief Title: A Phase Ib Study to Evaluate the Safety, Efficacy, and Pharmacokinetics of Cibisatamab in Combination With Atezolizumab After Pretreatment With Obinutuzumab in Participants With Previously Treated Metastatic Colorectal Adenocarcinoma
Status: Terminated | Phase: Phase 1 | Type: Interventional
Why Stopped: The Sponsor terminated the study because development of cibisatamab has been discontinued.
Sponsor: Hoffmann-La Roche (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: CO40939; 2018-003198-93 (EudraCT Number)
Record Dates: First submitted 2019-03-06; First posted 2019-03-07 (Actual); Last update posted 2024-08-09 (Actual); Status verified 2024-08

CONDITIONS: Colorectal Cancer
MeSH Terms: conditions — Colorectal Neoplasms | interventions — obinutuzumab; atezolizumab; cibisatamab; tocilizumab

STUDY DESIGN:
Oversight: FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (1):
- Obinutuzumab Pretreatment (OpT) + Cibisatamab + Atezolizumab (Experimental): Participants will receive obinutuzumab approximately 2 weeks before receiving atezolizumab and cibisatamab on Day 1 of each treatment cycle (cycle = 21 days).
  Interventions: Drug: Obinutuzumab; Drug: Atezolizumab; Drug: Cibisatamab; Drug: Tocilizumab

INTERVENTIONS:
Drug: Obinutuzumab — Obinutuzumab will be administered by intravenous (IV) infusion as either a split or single dose approximately 2 weeks before Cycle 1, Day 1 (cycle = 21 days).
  Other Names: Gazyva/Gazyvaro
Drug: Atezolizumab — Atezolizumab will be administered at a fixed dose of 1200 mg by IV infusion on Day 1 of each 21-day cycle until radiographic progression, unacceptable toxicity, or loss of clinical benefit.
  Other Names: Tecentriq
Drug: Cibisatamab — Cibisatamab will be administered at a fixed dose of 100 mg by IV infusion on Day 1 of each 21-day cycle until radiographic progression, unacceptable toxicity, or loss of clinical benefit.
Drug: Tocilizumab — Tocilizumab will be administered by IV infusion as necessary to manage adverse events (AEs)

SUMMARY:
CO40939 is a Phase Ib, open-label, multicenter, single-arm study designed to evaluate the safety, efficacy, pharmacokinetics, and immunogenicity of cibisatamab in combination with atezolizumab administered after pretreatment with obinutuzumab in patients with Stage IV microsatellite stable (MSS) metastatic colorectal cancer (mCRC) whose tumors have high carcinoembryonic antigen-related cell adhesion molecule 5 (CEACAM5) expression and who have progressed on two or more chemotherapy regimens. The study is composed of a safety run-in and an exploratory part.

ELIGIBILITY:
Inclusion criteria

* Histologically confirmed adenocarcinoma originating from the colon or rectum
* Metastatic disease not amenable to local treatment
* Tumors that are microsatellite stable or microsatellite instability low, as determined by a local, certified laboratory
* Tumors that have high carcinoembryonic antigen-related cell adhesion molecule 5 (CEACAM5) expression as determined by quantitative reverse transcription polymerase chain reaction (qRT-PCR) in an archival tumor sample or a fresh tumor biopsy and documented through central testing of a representative tumor tissue specimen performed at baseline
* Experienced disease progression during or within 3 months following the last administration of approved standard therapies
* Eastern Cooperative Oncology Group Performance Status of 0 or 1
* Life expectancy of >= 12 weeks
* Adequate hematologic and end-organ function
* Negative HIV test at screening
* Negative hepatitis B surface antigen test and total hepatitis B core antibody (HBcAb) test at screening, or positive total HBcAb test followed by a negative hepatitis B virus (HBV) DNA test at screening
* Negative hepatitis C virus (HCV) antibody test at screening, or positive HCV antibody test followed by a negative HCV RNA test at screening
* Negative human T-cell lymphotropic virus type 1 test for participants from endemic countries (Japan, countries in the Caribbean basin, South America, Central America, sub-Saharan Africa, and Malaysia)
* For women of childbearing potential: agreement to remain abstinent or use contraceptive methods, agreement to regular pregnancy testing, and agreement to refrain from donating eggs, women must remain abstinent or use contraceptive methods with a failure rate of < 1% per year during the treatment period and for 5 months after the final dose of atezolizumab, for 4 months after the final dose of cibisatamab, for 18 months after the final dose of obinutuzumab, and for 3 months after the final dose of tocilizumab
* For men: agreement to remain abstinent or use a condom, and agreement to refrain from donating sperm, with a female partner of childbearing potential or pregnant female partner, men must remain abstinent or use a condom during the treatment period and for 3 months after the final dose of cibisatamab, for 3 months after the final dose of obinutuzumab, and for 2 months after the final dose of tocilizumab to avoid exposing the embryo
* Lactic acid dehydrogenase (LDH) </= 2.5 x upper limit of normal (ULN)

Additional Inclusion Criteria for patient enrollment into Part 2 of the study:

- No prior treatment with regorafenib or Trifluridine/Tipiracil (TAS-102)

Exclusion criteria

* Symptomatic, untreated, or actively progressing central nervous system metastases
* Non-irradiated tumor lesions > 2 cm at critical sites where tumor swelling induced by cibisatamab is expected to lead to significant complications
* Dyspnea or peripheral capillary oxygen saturation < 92% at rest at baseline for patients with bilateral lung lesions or metastases in the remaining lung following lobectomy or pneumonectomy
* Spinal cord compression not definitively treated with surgery and/or radiation or previously diagnosed and treated spinal cord compression without evidence that disease has been clinically stable for >= 2 weeks prior to initiation of study treatment
* History of leptomeningeal disease and progressive multifocal leukoencephalopathy
* Uncontrolled tumor-related pain and pleural effusion or ascites requiring recurrent drainage procedures
* Participants with pericardial effusion
* Uncontrolled or symptomatic hypercalcemia
* Active or history of autoimmune disease or immune deficiency
* History of idiopathic pulmonary fibrosis, organizing pneumonia, drug-induced pneumonitis, or idiopathic pneumonitis, or evidence of active pneumonitis on screening chest computed tomography scan
* Active tuberculosis that has required treatment within 3 years prior initiation of study treatment or latent tuberculosis that has not been appropriately treated
* Uncontrolled hypertension, unstable angina, congestive heart failure of any New York Heart Association Class II or greater, serious cardiac arrhythmia requiring treatment and history of myocardial infarction within 6 months prior to initiation of study treatment
* Major surgical procedure, other than for diagnosis, within 4 weeks prior to initiation of study treatment, or anticipation of need for a major surgical procedure during the study
* History of malignancy other than CRC within 5 years prior to screening, with the exception of malignancies with a negligible risk of metastasis or death, such as adequately treated carcinoma in situ of the cervix, non-melanoma skin carcinoma, localized prostate cancer, ductal carcinoma in situ, or Stage I uterine cancer
* Known active infection, or reactivation of a latent infection, whether bacterial, viral, fungal, mycobacterial, or other pathogens, or any major episode of infection requiring hospitalization or treatment with IV antibiotics
* Prior allogeneic stem cell or solid organ transplantation
* Any other disease, metabolic dysfunction, physical examination finding, or clinical laboratory finding that contraindicates the use of an investigational drug, may affect the interpretation of the results, or may render the patient at high risk from treatment complications
* Treatment with a live, attenuated vaccine within 4 weeks prior to initiation of study treatment, or anticipation of need for such a vaccine during study treatment or within 5 months after the final dose of atezolizumab
* Current treatment with anti-viral therapy for HBV
* Treatment with any systemic anti-cancer therapy, including chemotherapy or hormonal therapy, within 28 days prior to initiation of study treatment
* Treatment with investigational therapy within 28 days prior to initiation of study treatment
* Prior treatment with any of the protocol-specified study treatments
* Prior treatment with T-cell bispecifics (TCBs), including CEACAM5-TCB, CD137 agonists or immune checkpoint blockade therapies, including anti-CTLA-4, anti-PD-1, and anti-PD-L1 therapeutic antibodies
* Treatment with systemic immunostimulatory agents within 4 weeks or 5 half-lives of the drug prior to initiation of study treatment
* Treatment with systemic immunosuppressive medication within 2 weeks prior to initiation of study treatment, or anticipation of need for systemic immunosuppressive medication during study treatment
* Adverse events from prior anti-cancer therapy that have not resolved to Grade 1 or better with the exception of alopecia of any grade and Grade <= 2 peripheral neuropathy
* History of severe allergic anaphylactic reactions to chimeric or humanized antibodies or fusion proteins
* Known hypersensitivity to Chinese hamster ovary cell products
* Known allergy or hypersensitivity to any of the study drugs or any of their excipients
* Pregnancy or breastfeeding, or intention of becoming pregnant during study treatment or within 5 months after the final dose of atezolizumab, within 4 months after the final dose of cibisatamab, within 18 months after the final dose of obinutuzumab, and within 3 months after the final dose of tocilizumab
* Participants with pleural effusion requiring drainage procedures
* Participants with pleural effusion and/or pleural lesions involving both lungs (i.e. bilateral pleural effusions; unliateral pleural effusion with pleural lesion in the contralateral lung)
* Participants with >10 bilateral pulmonary lesions (i.e. at least one lesion in each lung and more than 10 lung lesions in total)
* Participants with pulmonary miliary metastatic pattern (innumerable small lesions) or pulmonary lymphangitic carcinomatosis

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 47 (Actual)
Dates: Start 2019-05-07 (Actual); Primary Completion 2024-03-13 (Actual); Study Completion 2024-03-13 (Actual)

PRIMARY OUTCOMES:
Percentage of Participants with Adverse Events (AEs) | Up to 5 years
Confirmed Objective Response Rate (ORR) | Baseline up to 5 years

SECONDARY OUTCOMES:
Confirmed ORR, as Determined by an Independent Review Facility (IRF) According to Response Evaluation in Solid Tumors version 1.1 (RECIST v1.1) | Up to 5 years
Duration of Response (DOR) | From the first occurrence of a documented objective response to disease progression or death from any cause, whichever occurs first (up to 5 years)
Disease Control Rate (DCR) | Up to 5 years
Progression Free Survival (PFS) | From enrollment to the first occurrence of disease progression or death from any cause, whichever occurs first (up to 5 years)
Overall Survival (OS) | From enrollment to death from any cause (up to 5 years)
Total Clearance (CL) for Cibisatamab | At pre-defined intervals from Day 1 to progressive disease and/or treatment discontinuation (up to 5 years)
Volume of Distribution at Steady State (Vss) of Cibisatamab | At pre-defined intervals from Day 1 to progressive disease and/or treatment discontinuation (up to 5 years)
Area Under the Concentration-Time Curve (AUC0-t) for Cibisatamab | At pre-defined intervals from Day 1 to progressive disease and/or treatment discontinuation (up to 5 years)
Maximum Serum Concentration (Cmax) of Cibisatamab | At pre-defined intervals from Day 1 to progressive disease and/or treatment discontinuation (up to 5 years)
CL of Atezolizumab | At pre-defined intervals from Day 1, Cycle 1 through Cycle 8 (cycle = 21 days)
Vss of Atezolizumab | At pre-defined intervals from Day 1, Cycle 1 through Cycle 8 (cycle = 21 days)
AUC0-t of Atezolizumab | At pre-defined intervals from Day 1, Cycle 1 through Cycle 8 (cycle = 21 days)
Cmax of Atezolizumab | At pre-defined intervals from Day 1, Cycle 1 through Cycle 8 (cycle = 21 days)
CL of Obinutuzumab | At pre-defined intervals from the start of obinutuzumab pretreatment through Cycle 8 (cycle = 21 days)
Vss of Obinutuzumab | At pre-defined intervals from the start of obinutuzumab pretreatment through Cycle 8 (cycle = 21 days)
AUC0-t of Obinutuzumab | At pre-defined intervals from the start of obinutuzumab pretreatment through Cycle 8 (cycle = 21 days)
Cmax of Obinutuzumab | At pre-defined intervals from the start of obinutuzumab pretreatment through Cycle 8 (cycle = 21 days)
Incidence of Anti-Drug Antibodies (ADAs) to Cibisatamab | Baseline up to 5 years
Incidence of ADAs to Atezolizumab | Baseline up to 5 years
Incidence of ADAs to Obinutuzumab | Baseline up to 5 years

CONTACTS AND LOCATIONS:
Overall Officials: Clinical Trials, Study Director — Hoffmann-La Roche
Locations (13):
- United States (7):
  - Cedars Sinai Medical Center, Los Angeles, California
  - UCLA Cancer Center, Santa Monica, California
  - Stanford Comprehensive Cancer Center, Stanford, California
  - Yale University, New Haven, Connecticut
  - Memorial Sloan-Kettering Cancer Center, New York, New York
  - Duke Cancer Center, Durham, North Carolina
  - MD Anderson Cancer Center, Houston, Texas
- Rigshospitalet; Fase 1 Enhed - Onkologi, København Ø, Denmark
- France (2):
  - Centre Leon Berard; Departement Oncologie Medicale, Lyon
  - Institut Gustave Roussy, Villejuif
- Spain (3):
  - Hospital Univ Vall d'Hebron; Servicio de Oncologia, Sant Andreu de la Barca, Barcelona
  - Clinica Universitaria de Navarra; Servicio de Oncologia, Pamplona, Navarre
  - START Madrid-FJD, Hospital Fundacion Jimenez Diaz, Madrid

IPD SHARING:
Plan to Share IPD: Yes
Qualified researchers may request access to individual patient level data through the clinical study data request platform (www.vivli.org). Further details on Roche's criteria for eligible studies are available here (https://vivli.org/ourmember/roche/). For further details on Roche's Global Policy on the Sharing of Clinical Information and how to request access to related clinical study documents, see here (https://www.roche.com/research_and_development/who_we_are_how_we_work/clinical_trials/our_commitment_to_data_sharing.htm).